CLINICAL TRIAL: NCT06205914
Title: Management Of Patellar Fractures By Craniofacial Mesh Plate Osteosynthesis Augmented by Screws
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ayman Atef Ahmed, Resident-Orthopedic surgery depatement-Sohag university hospital, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Soh-Med-23-12-11MS
Record Dates: First submitted 2024-01-04; First posted 2024-01-16 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Patella Fracture
MeSH Terms: conditions — Patella Fracture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patient group (Experimental): patients more than 16 years old with patella frature
  Interventions: Procedure: fixation of patella fractures by craniofacial mesh plate osteosynthesis augmented by screws

INTERVENTIONS:
Procedure: fixation of patella fractures by craniofacial mesh plate osteosynthesis augmented by screws — patellar fracture fixation using MatrixNEURO Contourable Mesh plates (Synthes®). Made of titanium with an incredibly low profile
  Other Names: patella plate

SUMMARY:
Patellar fractures are challenging orthopedic injuries. Fractures that result in disruption of the extensor mechanism led to significant functional deficits. The goals of treatment for patella fractures include restoration of articular congruity, painless full range of motion of the knee, and recovery of extensor mechanism function.

The biomechanical construct chosen to fix patellar fractures is very important because of the subcutaneous location of the patella and the high level of force transmission that occurs through the patella during flexion and extension of the knee. Some studies have shown that during specific actions like walking or climbing downhill, the patella can see forces as high as 3200 N, equaling four to five times the standard body weight of a person. Achieving biomechanical stability during patellar fracture fixation is imperative as the stability of fixation is tested thousands of times as the knee is put through numerous cycles of flexion and extension during the recovery period. While tension band wiring with or without -K- wire, screw, or cerclage wire augmentation the most widely accepted form of treatment for patellar fractures, plate osteosynthesis is gaining popularity for certain fracture patterns. We present below a novel form of patellar fracture fixation using MatrixNEURO Contourable Mesh plates (Synthes®). Made of titanium with an incredibly low profile, these plates were initially designed for use in midface and craniofacial skeletal trauma.

However, we found that using these plates in treatment of patellar fractures has allowed stable fixation of complex, severely comminuted injuries The benefit of plate is adequate and stable reduction and maintenance of this reduction

ELIGIBILITY:
Inclusion Criteria:

patient with simple patella fractues more than 16 years.

Exclusion Criteria:

* Open fractures
* Preexisting deformity
* Ipsilateral femoral injuries

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
adequate and stable reduction | 1 year
  Evaluation of results of fixation of patellar fractures by craniofacial mesh plate

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

REFERENCES:
- [Background] Gwinner C, Mardian S, Schwabe P, Schaser KD, Krapohl BD, Jung TM. Current concepts review: Fractures of the patella. GMS Interdiscip Plast Reconstr Surg DGPW. 2016 Jan 18;5:Doc01. doi: 10.3205/iprs000080. eCollection 2016. PMID 26816667
- [Background] Benjamin J, Bried J, Dohm M, McMurtry M. Biomechanical evaluation of various forms of fixation of transverse patellar fractures. J Orthop Trauma. 1987;1(3):219-22. doi: 10.1097/00005131-198701030-00004. PMID 3506054
- [Background] Siljander M, Koueiter DM, Gandhi S, Wiater BP, Wiater PJ. Outcomes Following Low-Profile Mesh Plate Osteosynthesis of Patella Fractures. J Knee Surg. 2018 Oct;31(9):919-926. doi: 10.1055/s-0038-1625958. Epub 2018 Jan 30. PMID 29381883
- [Background] Volgas D, Dreger TK. The Use of Mesh Plates for Difficult Fractures of the Patella. J Knee Surg. 2017 Mar;30(3):200-203. doi: 10.1055/s-0037-1598078. Epub 2017 Feb 13. PMID 28192827